CLINICAL TRIAL: NCT00913484
Title: Disulfiram for Cocaine Abuse in Buprenorphine Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1R01DA012979 (NIH); 1R01DA012979 (NIH)
Record Dates: First submitted 2009-06-03; First posted 2009-06-04 (Estimated); Last update posted 2020-11-19 (Actual); Status verified 2020-11

CONDITIONS: Cocaine Dependence; Opioid Dependency
Keywords: Disulfiram; Buprenorphine; Cocaine dependence; Opioid dependence; Dopamine-Beta-Hydroxylase
MeSH Terms: conditions — Cocaine-Related Disorders; Opioid-Related Disorders | interventions — Disulfiram

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Disulfiram (Experimental): Disulfiram 250 mg per day
  Interventions: Drug: Disulfiram
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Disulfiram — Disulfiram 250 mg per day
  Arms: Disulfiram
Drug: Placebo — Placebo daily
  Arms: Placebo

SUMMARY:
The investigators are proposing a placebo-controlled clinical trial to evaluate the efficacy and potential mechanisms of action of disulfiram (versus placebo) for treating cocaine abuse in subjects with concurrent opiate dependence and cocaine abuse or dependence maintained on buprenorphine/naloxone combination.

DETAILED DESCRIPTION:
The Specific Aims and hypotheses for the proposed study are as follows:

1. To compare the efficacy of disulfiram versus placebo for the treatment of buprenorphine maintained patients with concurrent opioid and cocaine dependence. Study hypothesis 1 is that disulfiram is superior to placebo.
2. To evaluate whether dopamine-B-hydroxylase (DBH) genotypes associated with high, intermediate or low enzyme activity predict responses to disulfiram treatment of cocaine use in buprenorphine treated subjects. Study hypothesis 2 is that disulfiram efficacy is higher in subjects with low DBH compared to subjects with high DBH.
3. To explore whether baseline measures of alcohol use predict response to disulfiram. Study Hypothesis 3 is that the effects of disulfiram on cocaine use are independent of the severity of baseline alcohol use.

ELIGIBILITY:
Inclusion Criteria:

* English speaking adults ages 18 - 45.
* Meeting FDA criteria for agonist maintenance treatment and DSM-IV criteria for opioid dependence and cocaine dependence or abuse as assessed by SCID interview and documented by opioid positive and cocaine positive urine toxicology testing.
* Women of childbearing age will be included provided they agree to adequate contraception and to monthly pregnancy testing during the course of the study.

Exclusion Criteria:

* Current physiologic dependence on benzodiazepines or alcohol, unless first detoxified. Subjects who use/abuse alcohol will be included but will be cautioned about alcohol use during the study because of the possibility of an alcohol-disulfiram reaction.
* Use of the antibiotic agents metronidazole or clotrimazole, which have disulfiram-like effects in combination with alcohol.
* Presence of significant cardiovascular, renal, hepatic or neurologic illness. Subjects with markedly abnormal liver function tests (i.e., AST of ALT > 3X normal) will also be excluded.
* Presence of any of the following cardiovascular risk factors:

  * age > 45 years
  * history of cocaine-related chest pain
  * systolic blood pressure > 140 or diastolic blood pressure > 90
  * evidence of ischemia or past myocardial infarction on EKG
  * significant family history of risk (first degree relative with myocardial infarction prior to age 60)
  * elevated cholesterol (> 300 mg/dl), elevated LDL (> 170 mg/dl) or low HDL (< 20 mg/dl)
* Maintenance on methadone at doses greater than 30mg daily. Admittance to the study will only be offered to individuals who have been maintained on 30 mg of methadone or less daily for seven days prior to entering the study.
* Current suicide or homicide risk or current psychotic disorder.
* Inability to read or understand the symptom checklists.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 177 (Actual)
Dates: Start 2000-10; Primary Completion 2004-02 (Actual); Study Completion 2004-02 (Actual)

PRIMARY OUTCOMES:
Cocaine abstinence | 12 weeks

SECONDARY OUTCOMES:
Opioid abstinence | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Richard S. Schottenfeld, M.D., Principal Investigator — Yale University
Locations (2):
- United States (2):
  - The APT Foundation MRU, New Haven, Connecticut
  - Yale University School of Medicine, New Haven, Connecticut